CLINICAL TRIAL: NCT00049231
Title: Evaluation of Hypoxia by EF5 (NSC#684681) Binding in Cervix Cancer
Brief Title: EF5 to Detect Tumor Hypoxia in Patients With Stage IIB, Stage IIIB, or Stage IVA Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000258053; GOG-8002
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Cervical Cancer
Keywords: cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Immunohistochemistry; Biopsy

INTERVENTIONS:
Drug: EF5
Other: immunohistochemistry staining method
Procedure: biopsy

SUMMARY:
RATIONALE: Knowing the level of oxygen in tumor tissue may help predict the effectiveness of anticancer therapy. EF5 may be effective in measuring oxygen in tumor tissue and helping to predict the effectiveness of anticancer therapy.

PURPOSE: Diagnostic trial to study the effectiveness of EF5 in detecting tumor hypoxia in patients who have stage IIB, stage IIIB, or stage IVA cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relationship between the level of EF5 binding and pretreatment hemoglobin level, tumor size, and stage of disease in patients with stage IIB, IIIB, or IVA cervical cancer.
* Determine whether pretreatment tumor hypoxia (measured by EF5 binding) is associated with overall survival, progression-free interval, and local control in these patients.
* Determine the relationship between EF5 binding and CD-31 labeling (tumor vasculature) and Ki-67 labeling (cellular proliferation) in these patients.

OUTLINE: This is a multicenter study.

Patients receive EF5 IV over 1-2.5 hours on day 1. Tumor hypoxia is measured using immunohistochemical techniques. Biopsies are collected 1-2 days later. Blood is collected before EF5 is administered and again at the time of surgery.

Patients are followed approximately 1 month after surgery.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix

  * Stage IIB, IIIB, or IVA
  * Primary disease
* No prior treatment
* Must be enrolled on GOG-0191 protocol

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-3

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Alkaline phosphatase no greater than 3 times normal
* Hemoglobin less than 13 g/dL

Renal

* Creatinine no greater than 2 mg/dL

Cardiovascular

* No cardiac disease that would preclude safe administration of necessary fluid volumes

Pulmonary

* No chronic pulmonary disease that would preclude safe administration of necessary fluid volumes

Other

* No history of grade 3 or 4 peripheral neuropathy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must weigh no more than 180 kg

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gillian M. Thomas, BSc, MD, FRCPC, FRCR (Hon), Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (5):
- United States (5):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Colorado Gynecologic Oncology Group P.C., Denver, Colorado
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma